CLINICAL TRIAL: NCT01806363
Title: A Phase I Clinical Trial to Evaluate the Pharmacokinetic Interactions and Safety Between Telmisartan and Chlorthalidone in Healthy Male Volunteers.
Brief Title: Pharmacokinetic Interactions and Safety Study of Telmisartan and Chlorthalidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTECHL12I_1
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
Keywords: Pharmacokinetics; Safety; Male
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A: Telmisartan, Chlorthalidone + Telmisartan (Active Comparator): telmisartan 80mg : multiple dose administered orally chlorthalidone 25mg : multiple dose administered orally
  Interventions: Drug: Telmisartan 80mg; Drug: Chlorthalidone 25mg
- Part B: Chlorthalidone, Chlorthalidone + Telmisartan (Active Comparator): telmisartan 80mg : multiple dose administered orally chlorthalidone 25mg : multiple dose administered orally
  Interventions: Drug: Telmisartan 80mg; Drug: Chlorthalidone 25mg

INTERVENTIONS:
Drug: Telmisartan 80mg
Drug: Chlorthalidone 25mg

SUMMARY:
Clinical trial to evaluate the pharmacokinetic interactions and safety between telmisartan and chlorthalidone.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects
2. Age(yr)between 20 and 50
3. Signed written informed consent

Exclusion Criteria:

1. Known hypersensitivity to investigator product, thiazide, sulphonamide and other drugs or additive.
2. History of any siginificant Sickness, Cardiovascular, Respiratory, Renal, Endocrine, Neurological, Psychic, Cancer, Gasstrointestinal, Hematologic.
3. History of drug and/or alcohol abuse
4. Over 10 tobaccos a day
5. Other condition which in the opinion of the investigator preclude enrollment into the study

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Part A : AUC, Cmax of Telmisartan | Over a 24-hour sampling period
Part B : AUC, Cmax of Chlorthalidone | Over a 24-hour sampling period

SECONDARY OUTCOMES:
Part A : Cmin, tmax, CL/F of Telmisartan | Over a 24-hour sampling period
Part B : Cmin, tmax, CL/F of Chlorthalidone | Over a 24-hour sampling period

CONTACTS AND LOCATIONS:
Overall Officials: Young Ran Yoon, Associate Professor, Principal Investigator — KYUNGPOOK NATIONAL UNIVERSITY HOSPITAL, CLINICAL TRIAL CENTER
Locations (1):
- Kyungpook national university hospital Clionical center, Daegu, Gyeongsangbuk-do, South Korea

REFERENCES:
- [Derived] Seong SJ, Lim MS, Lee J, Ohk B, Gwon MR, Kim BK, Kim HJ, Yang DH, Lee HW, Kang WY, Yoon YR. Evaluation of a Pharmacokinetic Interaction between Telmisartan and Chlorthalidone in Healthy Male Adult Subjects. Clin Drug Investig. 2016 Aug;36(8):613-23. doi: 10.1007/s40261-016-0406-y. PMID 27206575